CLINICAL TRIAL: NCT03109457
Title: Hepatitis C Virus Detection in Oral Squamous Cell Carcinoma. (Retrospective-cohort Study)
Brief Title: Hepatitis C Virus Detection in Oral Squamous Cell Carcinoma
Status: Completed | Type: Observational
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Noura Kamal Aly, assistant lecturer, Oral and Maxillofacial pathology, Cairo University
Other Study IDs: CEBD-CU-2017-04-01
Record Dates: First submitted 2017-04-03; First posted 2017-04-12 (Actual); Last update posted 2020-02-05 (Actual); Status verified 2020-02

CONDITIONS: Hepatitis C
Keywords: Hepatitis C Virus; Oral squamous cell carcinoma
MeSH Terms: conditions — Hepatitis C; Squamous Cell Carcinoma of Head and Neck

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Oral squamous cell carcinoma: Sections (4-5 microns thick) will be cut for the immunohistochemical procedure, from each paraffin block and placed on positively charged (Opti-plus) slides by the technicians in the Oral and Maxillofacial laboratory setting.
  Hep C cAg : sc-58144, santa cruz biotechnology, USA) a mouse monoclonal antibody raised against Hepatitis C virus will be purchased and used for immunohistochemical staining.
  Interventions: Other: oral squamous cell carcinoma
- Control: Sections (4-5 microns thick) will be cut for the immunohistochemical procedure, from each paraffin block and placed on positively charged (Opti-plus) slides by the technicians in the Oral and Maxillofacial laboratory setting.
  Hep C cAg : sc-58144, santa cruz biotechnology, USA) a mouse monoclonal antibody raised against Hepatitis C virus will be purchased and used for immunohistochemical staining.
  Interventions: Other: oral squamous cell carcinoma

INTERVENTIONS:
Other: oral squamous cell carcinoma — Histological diagnosis of H&E stained sections will be performed according to WHO guidelines by 2 independent pathologists.
  Other Names: OSCC

SUMMARY:
Compare Hepatiis C Virus (HCV) detection between oral squamous cell carcinoma (OSCC) and normal tissues, to determine the possible relationship between HCV and OSCC.

DETAILED DESCRIPTION:
Patient / Population: Paraffin embedded tissue samples of OSCC. Indicator: OSCC patients Control: Normal patients Formalin fixed paraffin embedded specimens from blocks retrieved from the archives of the Oral and Maxillofacial Pathology Department, Faculty of dentistry, Kasr Alini hospital setting from January 2014 till February 2018. All clinical and histopathological data from medical reports, will be reviewed and data will be collected regarding age, sex, tumor location, history of smoking and alcohol consumption, nodal status, tumor recurrences and histological classification of the patients. The specimens will be obtained from 2 groups:-

1. OSCC specimens. Histological diagnosis of H&E stained sections will be performed according to World health organisation (WHO) guidelines by 2 independent pathologists.
2. Normal oral mucosa specimens (control).

outcome: I) Immunohistochemical detection of Hepatitis C core antigen (Hep C cAg) : sc-58144, santa cruz biotechnology, USA) a mouse monoclonal antibody raised against Hepatitis C virus will be purchased and used for immunohistochemical staining. Staining procedure using an automated system Ventana Benchmark. The four µm thick paraffin embedded tissue sections will be deparaffinized in three changes of xylene then microwaved for antigen retrieval. The slides will be incubated with primary antibody overnight in the humidity chamber at room temperature. Then, the slides will be incubated with secondary antibody. The peroxidase activity will be made visible with diaminobenzidine. Finally, counterstaining will be obtained using Mayer's hematoxylin.

The immunostained sections will be examined using analyzer computer system (Germany).

ELIGIBILITY:
Inclusion Criteria:

1. Presence of sufficient paraffin-embedded tumor material;
2. Presence of oral cavity cancer (including oral tongue, floor of mouth, gingiva, lips, buccal mucosa)
3. Absence of recurrent head and neck cancer
4. Absence of previous oncologic therapy;
5. Histological-proven squamous cell carcinoma.

   -

   Exclusion Criteria:

   subjects with missing information on age or sex will be excluded.

   -

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Formalin fixed paraffin embedded specimens from blocks retrieved from the archives of the Oral and Maxillofacial Pathology Department, Faculty of dentistry, Kasr Alini hospital setting from January 2014 till February 2018. All clinical and histopathological data from medical reports, will be reviewed and data will be collected regarding age, sex, tumor location, history of smoking and alcohol consumption, nodal status, tumor recurrences and histological classification of the patients
Sampling Method: Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2017-09-06 (Actual); Primary Completion 2018-02-07 (Actual); Study Completion 2018-09-15 (Actual)

PRIMARY OUTCOMES:
Hep C cAg by Immunohistochemistry | 5 years
  Hepatitis C core antigen by immunohistochemical analysis

CONTACTS AND LOCATIONS:
Overall Officials: Nora Ali, Msc, Principal Investigator — Assistant Lecturer at Oral and Maxillofacial pathology
Locations (1):
- Kasr ALini Hospital, Giza, Cairo Governorate, Egypt